CLINICAL TRIAL: NCT07124897
Title: The Effect of Virtual Reality-Supported Psychosocial Care on Psychosocial Health in Women Experiencing Perinatal Loss
Brief Title: Virtual Reality-Supported Psychosocial Care for Women After Perinatal Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu Dişli Çetinçay (Other)
Responsible Party: Sponsor-Investigator, Duygu Dişli Çetinçay, Lecturer, RN, MSc, PhD Student, Halic University
Organization: Halic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 30.01.2025-263
Record Dates: First submitted 2025-08-07; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Perinatal Death
Keywords: Virtual Reality; Perinatal Loss; Psychosocial; Nursing Care; Psychosocial Health
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial uses a parallel assignment model. Participants who meet the inclusion criteria are randomly assigned to one of two groups.
  The VR_PSYCARE group (experimental arm) receives VR-supported psychosocial nursing care based on Swanson's Theory of Caring, in addition to routine hospital care.
  The NONVR_PSYCARE group (control arm) receives psychosocial nursing care based on the Swanson's Theory of Caring, without VR, in addition to routine hospital care.
  The intervention consists of multiple phases: baseline assessment during hospitalization, face-to-face and at-home psychosocial care, and follow-up via telephone on Day 7 and Day 30 after discharge. Psychological outcomes-including depression, anxiety, stress, and grief-are measured using validated scales. Randomization ensures unbiased allocation, and the parallel design enables a direct comparison between the two intervention arms.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR_PSYCARE: VR-Supported Psychosocial Care + Routine Care (Experimental): Participants receive psychosocial nursing care based on Swanson's Theory of Caring, supported by VR, in addition to routine hospital care. The intervention includes face-to-face and at-home psychosocial care and telephone follow-up on Day 7 and Day 30 after discharge. VR content has two main components: (1) educational videos and multimedia materials addressing physical and reproductive health needs after perinatal loss, and (2) psychosocial content using 360° VR videos with guided breathing exercises, affirmations, and relaxation practices. This group is supported through follow-up calls and the continuation of at-home psychosocial care, including encouragement to practice breathing exercises, keep a daily journal, and receive supportive postpartum information.
  Interventions: Behavioral: VR-Supported Psychosocial Nursing Care Based on Swanson's Theory of Caring
- NONVR_PSYCARE: Psychosocial Care + Routine Care (Active Comparator): Participants receive psychosocial nursing care based on Swanson's Theory of Caring, without VR, in addition to routine hospital care. The intervention includes face-to-face and at-home psychosocial care and telephone follow-up on Day 7 and Day 30 after discharge. This group is supported through follow-up calls and the continuation of at-home psychosocial care, including encouragement to practice breathing exercises, keep a daily journal, and receive supportive postpartum information.
  Interventions: Behavioral: Psychosocial Nursing Care Based on Swanson's Theory of Caring

INTERVENTIONS:
Behavioral: VR-Supported Psychosocial Nursing Care Based on Swanson's Theory of Caring — This intervention involves psychosocial nursing care based on Swanson's Theory of Caring, supported by VR technology. It is applied to women experiencing perinatal loss, aiming to reduce grief, anxiety, depression, and stress, postpartum depression, and to enhance psychosocial well-being. The care is delivered face-to-face during hospitalization and includes emotional support, active listening, presence, and empathy, aligned with the core concepts of Swanson's theory. The VR component consists of immersive, calming 360-degree visual environments that are integrated into the care sessions to promote emotional regulation. The intervention continues with structured psychosocial support via telephone on day 7 and day 30 after discharge.
  Other Names: VR_PSYCARE; Swanson-Based VR Care
  Arms: VR_PSYCARE: VR-Supported Psychosocial Care + Routine Care
Behavioral: Psychosocial Nursing Care Based on Swanson's Theory of Caring — This intervention involves psychosocial nursing care based on Swanson's Theory of Caring, without the use of VR. It is delivered to women who have experienced perinatal loss, aiming to support emotional healing and reduce psychological symptoms such as grief, anxiety, depression, stress, and postpartum depression. The intervention is provided face-to-face during hospitalization and focuses on presence, listening, empathy, and emotional support in alignment with Swanson's caring processes. Follow-up support is also provided via telephone calls on day 7 and day 30 after discharge, continuing the psychosocial care process without any technological enhancement.
  Other Names: NONVR_PSYCARE; Swanson-Based Psychosocial Care
  Arms: NONVR_PSYCARE: Psychosocial Care + Routine Care

SUMMARY:
The goal of this clinical trial is to evaluate the effect of virtual reality (VR)-supported psychosocial nursing care on the psychosocial health of women aged 18 and older who have experienced perinatal loss (≥20 weeks of gestation).

The main questions it aims to answer are:

Does VR-supported psychosocial care reduce depression, anxiety, stress, perinatal grief, and postpartum depression compared to psychosocial care without VR support?

Researchers will compare two groups:

VR-supported psychosocial care Psychosocial care without VR support

Participants will complete baseline psychosocial assessments during hospital admission, receive psychosocial nursing care based on Swanson's Theory of Caring - with or without VR support - during hospitalization, take part in follow-up interviews on Day 7 and Day 30 after discharge, and continue the psychosocial care process at home, including practicing breathing exercises, keeping a daily journal, and receiving supportive information about coping after perinatal loss.

DETAILED DESCRIPTION:
Perinatal loss, typically resulting from miscarriage, stillbirth, or neonatal death, is defined as an unwanted pregnancy or infant loss. Considered a traumatic life event, perinatal loss affects the family beyond the loss of the baby, leading to feelings of hopelessness and disappointment about the future. It is a profound source of distress that can result in depression, anxiety, stress, grief, and postpartum depression.

Psychosocial nursing care for women during this period plays a critical role; however, innovative approaches are needed to enhance its effectiveness. Virtual reality (VR) technology provides an immersive environment that can promote relaxation, distract from distressing thoughts, and increase engagement in therapeutic activities. Integrating VR into psychosocial care may help address the complex emotional needs of women following perinatal loss.

This study will evaluate VR-supported psychosocial nursing care, based on Swanson's Theory of Caring, on the psychosocial health outcomes of women aged 18 years and older who have experienced perinatal loss. The intervention includes both educational content addressing physical and reproductive health needs and VR content designed to support psychosocial well-being (360° videos, e.g., forest, seaside), combined with voice-guided breathing exercises, affirmations, and guided relaxation practices.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Being 18 years of age or older
* Having access to a smartphone and the internet
* Having experienced a pregnancy loss at ≥20 weeks of gestation

Exclusion Criteria:

* Experiencing neonatal loss
* Having a diagnosed psychiatric disorder
* Having a visual or hearing impairment
* Becoming pregnant through infertility treatment
* Inability to speak or understand Turkish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety, and Stress Levels | Baseline (hospital admission), Day 7 post-discharge, Day 30 post-discharge
  The primary outcome measure will be assessed using the Depression Anxiety Stress Scale-21 (DASS-21), a shortened version of the original 42-item scale (DASS-42). The DASS-21 consists of 21 items grouped into three subscales: depression, anxiety, and stress, with each subscale comprising seven items. Responses are rated on a 4-point Likert scale, and total scores for each subscale are calculated by summing the item scores and multiplying the result by two. Higher scores indicate greater severity of symptoms. The scale will be administered at three time points: baseline (upon hospital admission), Day 7 post-discharge, and Day 30 post-discharge.
Perinatal Grief Levels | Baseline (hospital admission), Day 7 post-discharge, Day 30 post-discharge
  Perinatal grief will be assessed using the Perinatal Grief Scale - Short Form (PGS), developed to measure the intensity of grief following perinatal loss. The scale consists of 33 items in its original form; however, the short form includes 32 items rated on a 5-point Likert scale. It comprises three subscales: active grief, difficulty coping, and despair, each containing 11 items. Items are summed to provide a total score ranging from 32 to 160, with higher scores indicating greater levels of grief. Except for items 11 and 32, all items are reverse-scored. The scale can be administered within the first two weeks post-loss or during later stages. The PGS-SF will be administered at baseline (hospital admission), Day 7 post-discharge, and Day.
Postpartum Depression Levels | Day 7 post-discharge, Day 30 post-discharge
  Postpartum depression will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), developed to screen for the risk of depression in women during the postnatal period. The EPDS consists of 10 items rated on a 4-point Likert scale, with each item scored from 0 to 3. Total scores range from 0 to 30, with higher scores indicating greater risk of postpartum depression. Items 1, 2, and 4 are scored positively, while the remaining items are reverse-scored. A cutoff score of 13 is used; scores of 13 or higher indicate a potential risk for postpartum depression, while scores of 12 or lower suggest a lower risk. The scale will be administered at Day 7 and Day 30 post-discharge.

OTHER OUTCOMES:
Assessment of Sociodemographic, Obstetric, and Gynecological Characteristics | Baseline (hospital admission)
  A researcher-designed Participant Information Form will be used to collect key background information from participants. The form includes selected items on sociodemographic characteristics (e.g., age, education level), obstetric history (e.g., number of pregnancies, pregnancy planning), and gynecological features (e.g., previous pregnancy loss, complications). It was developed based on relevant literature and will be administered at baseline (hospital admission) to describe the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Dişli Çetinçay, RN, MSc, Principal Investigator — Haliç University
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the absence of participant consent for external data sharing and institutional policies that restrict the release of raw data.

REFERENCES:
- [Background] Chiu PL, Li H, Yap KY, Lam KC, Yip PR, Wong CL. Virtual Reality-Based Intervention to Reduce Preoperative Anxiety in Adults Undergoing Elective Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2340588. doi: 10.1001/jamanetworkopen.2023.40588. PMID 37906193
- [Background] Kersting A, Wagner B. Complicated grief after perinatal loss. Dialogues Clin Neurosci. 2012 Jun;14(2):187-94. doi: 10.31887/DCNS.2012.14.2/akersting. PMID 22754291
- [Background] Kalanlar B. Hospital Practices for Parents Following Perinatal Loss. Omega (Westport). 2020 Nov;82(1):92-104. doi: 10.1177/0030222818803809. Epub 2018 Oct 3. PMID 30282521
- [Background] Fenstermacher K, Hupcey JE. Perinatal bereavement: a principle-based concept analysis. J Adv Nurs. 2013 Nov;69(11):2389-400. doi: 10.1111/jan.12119. Epub 2013 Mar 4. PMID 23458030
- [Background] Mecdi Kaydirak M, Aslan E. Efficacy of Nursing Support in the Pre- and Postmedical Termination of Pregnancy Phases: A Randomized Study. Omega (Westport). 2021 Nov;84(1):51-68. doi: 10.1177/0030222819877791. Epub 2019 Sep 24. PMID 31550199
- [Background] Demirel G, Ertekin Pinar S, Bilgic D. Anxiety levels and methods of coping with stress of adolescents undergoing their first gynecological examination. J Psychosom Obstet Gynaecol. 2020 Jun;41(2):131-136. doi: 10.1080/0167482X.2019.1643314. Epub 2019 Jul 22. PMID 31328602
- [Background] Engindeniz, A. N., Küey, L., & Kültür, S. (1996). Edinburgh Doğum Sonrası Depresyon Ölçeği Türkçe Formu Geçerlilik ve Güvenilirlik Çalışması. Bahar Sempozyumları, 1, 51-52.
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Köneş, M. Ö., Mecdi Kaydirak, M., Aslan, E., & Yildiz, H. (2017). Perinatal Yas Ölçeği (33 maddeli Kısa Sürüm): Türkçe geçerlilik ve güvenilirlik çalışması. Anadolu Psikiyatri Dergisi, 18(3), 231-236. doi: 10.5455/apd.234509.
- [Background] Toedter LJ, Lasker JN, Janssen HJ. International comparison of studies using the perinatal grief scale: a decade of research on pregnancy loss. Death Stud. 2001 Apr-May;25(3):205-28. doi: 10.1080/07481180125971. PMID 11785540
- [Background] Sarıçam, H. (2018). The Psychometric Properties of Turkish Version of Depression Anxiety Stress Scale-21 (DASS-21) in Community and Clinical Samples. Journal of Cognitive-Behavioral Psychotherapy and Research, 7(1), 1.
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811